CLINICAL TRIAL: NCT03438396
Title: A Single Arm, Multicenter, International Trial of Tisotumab Vedotin (HuMax®-TF-ADC) in Previously Treated, Recurrent or Metastatic Cervical Cancer
Brief Title: A Trial of Tisotumab Vedotin in Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genmab (Industry); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Belgian Gynaecological Oncology Group (Other); Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1015-04; innovaTV 204 (Other: Genmab)
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tisotumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): tisotumab vedotin (IV), 2.0 mg/kg, every 3 weeks (1Q3W)
  Interventions: Drug: tisotumab vedotin

INTERVENTIONS:
Drug: tisotumab vedotin — All patients will be treated with tisotumab vedotin once every three weeks until progression or toxicity
  Other Names: TIVDAK

SUMMARY:
A Single arm, Multicenter, International Trial of Tisotumab Vedotin (HuMax®-TF-ADC) in Previously Treated, Recurrent or Metastatic Cervical Cancer.

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the efficacy and safety/tolerability of tisotumab vedotin in patients with previously treated, recurrent or metastatic cervical cancer. Tisotumab vedotin is an antibody-drug conjugate (ADC) targeting tissue factor (TF), a protein aberrantly expressed in a wide number of tumors including cervical cancer. Preliminary safety and efficacy data observed in a cohort of previously treated cervical cancer patients suggest a positive benefit risk profile for this population of high unmet need.

ELIGIBILITY:
Inclusion Criteria

* Patients with extra-pelvic metastatic or recurrent cervical cancer including squamous cell, adenocarcinoma or adenosquamous histology who have experienced disease progressed on standard of care chemotherapy in combination with bevacizumab, if eligible.
* Measurable disease according to RECIST v1.1 as assessed by IRC.
* Age ≥ 18 years.
* Acceptable renal function
* Acceptable liver function
* Acceptable hematological status
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A negative serum pregnancy test for patients of reproductive potential.
* All patients must provide a fresh or archival biopsy during screening.
* Following receipt of verbal and written information about the trial, patients must provide signed informed consent before any trial-related activity is carried out.

Exclusion Criteria

* Have received no more than 2 prior systemic treatment regimens for recurrent or metastatic cervical cancer.
* Known past or current coagulation defects leading to an increased risk of bleeding;
* Ongoing major bleeding
* Active ocular surface disease
* Known past or current malignancy other than the inclusion diagnosis.
* Peripheral neuropathy grade ≥ 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cervical cancer
Enrollment: 102 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Arizona Oncology Associate - Biltmore Cancer Center, Phoenix, Arizona
  - UCLA Dept. of OBGYN, Los Angeles, California
  - Southern Baptist Hospital of Florida, Inc, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Gynecologic Oncology, Atlanta, Georgia
  - Community Hospital East, Indianapolis, Indiana
  - Louisville Oncology, Louisville, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - MD Anderson Cancer Center at Cooper University Hospital, Camden, New Jersey
  - University of New Mexico Comprehensive Cancer Center (UNMCCC), Albuquerque, New Mexico
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Hilliard, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Abington Memorial Hospital, Willow Grove, Pennsylvania
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - UT Health McGovern Medical School, Houston, Texas
  - Froedtert & Medical College Clinics, Milwaukee, Wisconsin
- Belgium (10):
  - AZ Sint-Jan Brugge-Oostende av, Bruges
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Algemeen Ziekenhuis Maria MiddelaresMedical Oncology - IKG, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - UZLeuvenGynaecologische oncologie, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - CHC SAINT Montlegia, Liège
  - CHU de LIEGE/ Oncologie Médicale, domaine universitaire du Sart Tilman, Liège
  - CHU UCL Namur site de Sainte Elisabeth, Namur
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc Onkologic, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Na Bulovce, Gynekologicko-porodnicka kl, Prague
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
- Germany (3):
  - Kliniken Essen-Mitte, Düsseldorf
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Universität München, Münich
- Italy (5):
  - Policlinico S.Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna
  - Irst Irccs, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Naples
  - Policlinico Universitario Agostino Gemelli, UOC Patologia Ostetrica e Ginecologica, Rome
- Spain (8):
  - Hospital Teresa Herrera-CHUAC, A Coruña
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Duran I Reynals ICO Hospitalet, L'Hospitalet de Llobregat
  - Clínica Universidad de Navarra (Sede Madrid), Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Edificio dotacional de Oncología, Madrid
  - Fundacion Hospital Son Llatzer, Palma de Mallorca
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng S, Gunawan R, Passey C, Voellinger J, Polhamus D, Gerritsen A, O'Day C, Carret AS, Soumaoro I, Gupta M, Hanley WD. Exposure-safety Markov modeling of ocular adverse events in patient populations treated with tisotumab vedotin. J Pharmacokinet Pharmacodyn. 2025 Oct 3;52(5):55. doi: 10.1007/s10928-025-10003-w. PMID 41044356
- [Derived] Passey C, Voellinger J, Gibiansky L, Gunawan R, Nicacio L, Soumaoro I, Hanley WD, Winter H, Gupta M. Exposure-safety and exposure-efficacy analyses for tisotumab vedotin for patients with locally advanced or metastatic solid tumors. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1262-1273. doi: 10.1002/psp4.13007. Epub 2023 Jul 26. PMID 37496366
- [Derived] Coleman RL, Lorusso D, Gennigens C, Gonzalez-Martin A, Randall L, Cibula D, Lund B, Woelber L, Pignata S, Forget F, Redondo A, Vindelov SD, Chen M, Harris JR, Smith M, Nicacio LV, Teng MSL, Laenen A, Rangwala R, Manso L, Mirza M, Monk BJ, Vergote I; innovaTV 204/GOG-3023/ENGOT-cx6 Collaborators. Efficacy and safety of tisotumab vedotin in previously treated recurrent or metastatic cervical cancer (innovaTV 204/GOG-3023/ENGOT-cx6): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2021 May;22(5):609-619. doi: 10.1016/S1470-2045(21)00056-5. Epub 2021 Apr 9. PMID 33845034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Europe and the US.
Pre-assignment Details: A 102 participants with Recurrent or Metastatic Cervical Cancer were enrolled in the study and out of which 101 participants received study treatment. These participants were assessed until the participant experienced IRC-verified disease progression, started new anti-cancer therapy, discontinued the trial, or died.
Groups:
- Tisotumab Vedotin: Participants received IV tisotumab vedotin 2.0 mg/kg Q3W until radiographic disease progression verified by the IRC, unacceptable AEs requiring drug discontinuation, withdrawal of consent, lost to follow up or death, whichever occurred first.
Period: Overall Study
Arm/Group | Tisotumab Vedotin
Started | 102
Treated | 101
Completed | 0
Not Completed | 102
Not completed — Reason Not Specified | 9
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2
Not completed — Death | 85
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of tisotumab vedotin.
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.66 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 95
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response (OR) as Assessed by the Independent Review Committee (IRC)
Description: The confirmed OR is defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) based upon RECIST v1.1, assessed by the IRC. The CR is disappearance of all target and non-target lesions and no new lesions. A confirmed CR is 2 CRs (CR-CR sequence) that were separated by at least 4 weeks with no evidence of progression in-between. The PR is ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no unequivocal progression of existing non-target lesions and no new lesion. A confirmed PR is PR-PR sequence or PR-CR sequence that were separated by at least 4 weeks. The intermediate missing (Not Evaluable [NE]) scan evaluations between response scan and confirmation scan were allowed, eg, PR-NE-PR and PR-NE-NE-PR was considered PR confirmed (a repeat scan not earlier than 4 weeks after initial scan documenting response). 95% CI was calculated using the Clopper-Pearson method.
Time Frame: From Day 1 through IRC verified disease progression, initiation of new anticancer therapy, study withdrawal, or death, whichever occurred first (approximately 20 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Percentage of Participants | 23.8 [15.9 to 33.3]
Statistical Analysis 1: Comparison: Tisotumab Vedotin; Test type: Other — The statistical hypotheses was tested to address ORR <= 11% vs. ORR > 11%; p = 0.0002, one-sided exact test

2. Secondary Outcome: Duration of Response (DOR) as Assessed by the IRC
Description: The DOR is defined as the duration from the first documented response of CR or PR (the start date of response, not the date when response was confirmed) to the date of the first documented progression disease (PD) verified by IRC or death. Based upon RECIST v1.1, the CR is defined as disappearance of all target and non-target lesions and no new lesions; the PR is defined as ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no unequivocal progression of existing non-target lesions and no new lesion; and the PD is defined as at least 20% increase in the sum of diameters of target lesions (compared to baseline), unequivocal progression of existing non-target lesions, and/or new lesion. The DOR was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through IRC verified disease progression, initiation of new anticancer therapy, study withdrawal, or death, whichever occurred first (approximately 49 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin. The DOR was analyzed for those participants in FAS who achieved confirmed OR, as assessed by the IRC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 24
Months | 8.3 [4.2 to 13.5]

3. Secondary Outcome: Percentage of Participants With Confirmed OR as Assessed by the Investigator
Description: The confirmed OR is defined as best overall response of confirmed CR or confirmed PR based upon RECIST v1.1, assessed by the investigator. The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as 2 CRs (CR-CR sequence) that were separated by at least 4 weeks with no evidence of progression in-between. The PR is defined as ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no unequivocal progression of existing non-target lesions and no new lesion. A confirmed PR is defined as PR-PR sequence or PR-CR sequence that were separated by at least 4 weeks. The intermediate missing (NE) scan evaluations between the response scan and the confirmation scan were allowed, eg, PR-NE-PR and PR-NE-NE-PR was considered PR confirmed (a repeat scan not earlier than 4 weeks after initial scan documenting response). 95% CI was calculated using the Clopper-Pearson method.
Time Frame: From Day 1 through investigator verified disease progression, initiation of new anticancer therapy, study withdrawal, or death, whichever occurred first (approximately 49 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Percentage of Participants | 20.8 [13.4 to 30.0]

4. Secondary Outcome: DOR as Assessed by the Investigator
Description: The DOR is defined as the duration from the first documented response of CR or PR (the start date of response, not the date when response was confirmed) to the date of the first documented PD verified by investigator or death. Based upon RECIST v1.1, the CR is defined as disappearance of all target and non-target lesions and no new lesions; the PR is defined as ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no unequivocal progression of existing non-target lesions and no new lesion; and the PD is defined as at least 20% increase in the sum of diameters of target lesions (compared to baseline), unequivocal progression of existing non-target lesions, and/or new lesion. The DOR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin. The DOR was analyzed for those participants in FAS who achieved confirmed OR, as assessed by the investigator.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 21
Months | 8.2 [3.7 to 18.4]

5. Secondary Outcome: Time to Response (TTR) as Assessed by the IRC
Description: The TTR is defined as the duration from the start of study drug to the first documented response of either CR or PR based on RECIST v1.1, assessed by the IRC. A confirmed CR is defined as 2 CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as 2 PRs (≥ 30% decrease in the sum of diameters of target lesions compared to baseline and no unequivocal progression of existing non-target lesions and no new lesion) or an un-confirmed PR and an un-confirmed CR or achieved PR-NE-PR or PR-NE-NE-PR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 2
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin. The TTR was analyzed for those participants in FAS who achieved confirmed OR, as assessed by the IRC.
Measure: Median (Full Range); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 24
Months | 1.4 [1.1 to 5.1]

6. Secondary Outcome: TTR as Assessed by the Investigator
Description: The TTR is defined as the duration from the start of study drug to the first documented response of either CR or PR based on RECIST v1.1, assessed by the investigator. A confirmed CR is defined as 2 CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as 2 PRs (≥ 30% decrease in the sum of diameters of target lesions compared to baseline and no unequivocal progression of existing non-target lesions and no new lesion) or an un-confirmed PR and an un-confirmed CR or achieved PR-NE-PR or PR-NE-NE-PR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 3
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin. The TTR was analyzed for those participants in FAS who achieved confirmed OR, as assessed by the investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 21
Months | 1.4 [1.1 to 4.5]

7. Secondary Outcome: Progression Free Survival (PFS) as Assessed by the IRC
Description: The PFS is defined as the time from the start of study drug until the first documentation of PD based on RECIST v1.1, as assessed by the IRC or death due to any cause, whichever occurred first. The PD based upon RECIST v1.1 is defined as at least 20% increase in the sum of diameters of target lesions (compared to baseline), unequivocal progression of existing non-target lesions, and/or new lesion. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 2
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Months | 4.2 [3.0 to 4.4]

8. Secondary Outcome: PFS as Assessed by the Investigator
Description: The PFS is defined as the time from the start of study drug until the first documentation of PD based on RECIST v1.1, as assessed by the investigator or death due to any cause, whichever occurred first. The PD based upon RECIST v1.1 is defined as at least 20% increase in the sum of diameters of target lesions (compared to baseline), unequivocal progression of existing non-target lesions, and/or new lesion. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Months | 4.1 [3.3 to 4.6]

9. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 until death or withdrawal from the study, whichever occurred first (approximately 49 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Months | 12.3 [9.6 to 14.1]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE is defined as an AE that meets one of the following criteria: fatal or life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; medically significant (an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above [medical and scientific judgment must be exercised in deciding whether an AE is "medically important"]); required inpatient hospitalization or prolongation of existing hospitalization. A TEAE is defined as an AE occurring or worsening between the first dose of tisotumab vedotin and 30 days after the last dose received.
Time Frame: From Day 1 through 30 days after the last dose of study drug (approximately 49 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Participants
  Any TEAE | 101
  Any TESAE | 44

11. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Laboratory abnormalities that induced clinical signs or symptoms, required concomitant therapy or required changes during treatment emergent period were reported as TEAEs. Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Time Frame: From Day 1 through 30 days after the last dose of study drug (approximately 49 months)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
Participants
  Anaemia | 34
  Neutropenia | 4
  Iron deficiency anaemia | 3
  Leukocytosis | 1
  Leukopenia | 1
  Thrombocytopenia | 1
  Thrombocytosis | 1
  Hypokalaemia | 6
  Hypomagnesaemia | 6
  Hypocalcaemia | 4
  Hyperglycaemia | 3
  Hypercreatininaemia | 2
  Hyperuricaemia | 2
  Hypercalcaemia | 1
  Hypernatraemia | 1
  Hypoalbuminaemia | 1
  Hyponatraemia | 1
  Activated partial thromboplastin time prolonged | 3
  Neutrophil count decreased | 3
  Blood creatinine increased | 2
  C-reactive protein increased | 2
  International normalised ratio increased | 2
  Lymphocyte count decreased | 2
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Blood alkaline phosphatase increased | 1
  Blood bicarbonate decreased | 1
  Blood creatine phosphokinase increased | 2
  Blood potassium decreased | 1
  Creatinine renal clearance decreased | 1
  Platelet count decreased | 2
  Prothrombin time prolonged | 1
  White blood cell count decreased | 1
  Hyperthyroidism | 1
  Hypothyroidism | 1
  Hypertransaminasaemia | 3
  Hyperbilirubinaemia | 1
  Haematuria | 10

12. Secondary Outcome: Plasma Concentrations of Tisotumab Vedotin (HuMax-TF), Tisotumab Vedotin Antibody-drug Conjugate (HuMax-TF-ADC), and Free Monomethyl Auristatin E (MMAE)
Description: Plasma concentrations of HuMax-TF, HuMax-TF-ADC, and Free MMAE measures on Cycle 1 Day 1 (predose and end of infusion) and Cycle 6 Day 1 (predose and end of infusion) are reported.
Time Frame: Predose and end of infusion of Cycle 1 Day 1 (C1D1) and Cycle 6 Day 1 (C6D1)
Population: FAS included all participants who received at least 1 dose of tisotumab vedotin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 101
ng/mL
  HuMax-TF (C1D1-predose): number analyzed (Participants) | 98
  HuMax-TF (C1D1-predose) | 163.48 (60.70)
  HuMax-TF (C1D1-end of infusion): number analyzed (Participants) | 98
  HuMax-TF (C1D1-end of infusion) | 41691.0 (68.02)
  HuMax-TF (C6D1-predose): number analyzed (Participants) | 54
  HuMax-TF (C6D1-predose) | 150.0 (0.0)
  HuMax-TF (C6D1-end of infusion): number analyzed (Participants) | 54
  HuMax-TF (C6D1-end of infusion) | 36941 (25.88)
  HuMax-TF-ADC (C1D1-predose): number analyzed (Participants) | 97
  HuMax-TF-ADC (C1D1-predose) | 30.0 (0.0)
  HuMax-TF-ADC (C1D1-end of infusion): number analyzed (Participants) | 97
  HuMax-TF-ADC (C1D1-end of infusion) | 38105 (92.62)
  HuMax-TF-ADC (C6D1-predose): number analyzed (Participants) | 54
  HuMax-TF-ADC (C6D1-predose) | 30.0 (0.0)
  HuMax-TF-ADC (C6D1-end of infusion): number analyzed (Participants) | 53
  HuMax-TF-ADC (C6D1-end of infusion) | 36270.0 (28.29)
  MMAE (C1D1-predose): number analyzed (Participants) | 96
  MMAE (C1D1-predose) | 12.50 (0.0)
  MMAE (C1D1-end of infusion): number analyzed (Participants) | 97
  MMAE (C1D1-end of infusion) | 171.27 (102.05)
  MMAE (C6D1-predose): number analyzed (Participants) | 53
  MMAE (C6D1-predose) | 46.71 (146.11)
  MMAE (C6D1-end of infusion): number analyzed (Participants) | 54
  MMAE (C6D1-end of infusion) | 177.46 (82.62)

13. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to Tisotumab Vedotin
Description: Number of participants with positive ADA titer to tisotumab vedotin at baseline and post-baseline are reported. Baseline is defined as the latest available measurement made before the first dose of tisotumab vedotin. For post-baseline results, a participant was considered ADA positive if either ADA is negative at baseline and at least one post-baseline result is positive or positive at baseline and at least one positive post-baseline result with a titer higher than baseline.
Time Frame: Predose of each treatment cycle (Cycle 1 to 21) and end of treatment visit (approximately 49 months)
Population: Participants in FAS (received at least 1 dose of tisotumab vedotin) and who had ADA results at baseline and post-baseline are analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 93
Participants
  ADA positive at Baseline | 2
  ADA positive at post-baseline | 5

ADVERSE EVENTS:
Time Frame: From Day 1 through 30 days after the last dose of study drug (approximately 49 months)
Arm/Group | Tisotumab Vedotin
All-Cause Mortality (participants affected / at risk) | 86/101
Serious Adverse Events (participants affected / at risk) | 44/101
Other Adverse Events (participants affected / at risk) | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisotumab Vedotin (N=101)
Pneumonia (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Death (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
General physical condition abnormal (Investigations) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Ulcerative Keratitis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisotumab Vedotin (N=101)
Nausea (Gastrointestinal disorders) | 41 (51)
Diarrhoea (Gastrointestinal disorders) | 25 (29)
Constipation (Gastrointestinal disorders) | 20 (20)
Vomiting (Gastrointestinal disorders) | 17 (25)
Abdominal pain (Gastrointestinal disorders) | 13 (18)
Dry mouth (Gastrointestinal disorders) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 35 (47)
Asthenia (General disorders) | 18 (18)
Pyrexia (General disorders) | 15 (38)
Influenza like illness (General disorders) | 7 (7)
Oedema peripheral (General disorders) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 39 (39)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (18)
Rash (Skin and subcutaneous tissue disorders) | 14 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6)
Conjunctivitis (Infections and infestations) | 31 (49)
Urinary tract infection (Infections and infestations) | 10 (12)
Nasopharyngitis (Infections and infestations) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Dry eye (Eye disorders) | 25 (30)
Keratitis (Eye disorders) | 11 (15)
Blepharitis (Eye disorders) | 7 (10)
Punctate keratitis (Eye disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 (49)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (24)
Headache (Nervous system disorders) | 8 (12)
Anaemia (Blood and lymphatic system disorders) | 33 (39)
Decreased appetite (Metabolism and nutrition disorders) | 18 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6)
Weight decreased (Investigations) | 14 (14)
Haematuria (Renal and urinary disorders) | 9 (11)
Vaginal haemorrhage (Reproductive system and breast disorders) | 10 (13)
Insomnia (Psychiatric disorders) | 10 (10)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3)
Retching (Gastrointestinal disorders) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Subileus (Gastrointestinal disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 3 (4)
Facial pain (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion site coldness (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucosal disorder (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (2)
Parotitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3)
Stenotrophomonas infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Amblyopia (Eye disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Chalazion (Eye disorders) | 1 (1)
Conjunctival erosion (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (3)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vision blurred (Eye disorders) | 3 (3)
Ulcerative keratitis (Eye disorders) | 4 (4)
Trichiasis (Eye disorders) | 2 (2)
Retinal exudates (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 4 (4)
Noninfective conjunctivitis (Eye disorders) | 1 (1)
Meibomianitis (Eye disorders) | 3 (3)
Meibomian gland dysfunction (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 4 (4)
Keratopathy (Eye disorders) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 3 (3)
Entropion (Eye disorders) | 3 (3)
Corneal scar (Eye disorders) | 1 (1)
Corneal erosion (Eye disorders) | 2 (2)
Corneal bleeding (Eye disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3)
Sensory loss (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Paranasal sinus haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 2 (2)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 4 (6)
Neuralgia (Nervous system disorders) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 3 (4)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Burning sensation (Nervous system disorders) | 4 (4)
Weight increased (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 2 (2)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 5 (6)
Chromaturia (Renal and urinary disorders) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 4 (5)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Genital swelling (Reproductive system and breast disorders) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Allergy to metals (Immune system disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hot flush (Vascular disorders) | 5 (6)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1)
Radiation associated haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Conjunctival scar (Injury, poisoning and procedural complications) | 1 (1)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 12 months but less than 18 months from the end of study (database lock). The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT03438396/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT03438396/SAP_001.pdf